CLINICAL TRIAL: NCT05135650
Title: Pharmacokinetics of a SARS-CoV-2 Monoclonal Antibody in Hematopoietic Stem Cell Transplant Recipients (COVIDMAB)
Brief Title: Pharmacokinetics of Sotrovimab as Pre-exposure Prophylaxis for COVID-19 in Hematopoietic Stem Cell Transplant Recipients, COVIDMAB Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to FDA withdrawal of the emergency use authorization (EUA) for sotrovimab
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Marrow Donor Program (Other); Vir Biotechnology, Inc. (Industry)
Responsible Party: Principal Investigator, Alpana Waghmare, Assistant Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RG1121602; NCI-2021-05949 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10691 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-11-23; First posted 2021-11-26 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: COVID-19 Infection; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms | interventions — sotrovimab; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (Sotrovimab) (Experimental): Patients receive sotrovimab IV over 30 minutes within 1-7 days prior to the start of pre-transplant conditioning. Patients also undergo blood and nasal swab sample collection throughout the trial.
  Interventions: Other: Questionnaire Administration; Biological: Sotrovimab; Procedure: Biospecimen Collection

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Biological: Sotrovimab — Given IV
  Other Names: Anti-SARS-CoV-2 Spike Protein Monoclonal Antibody VIR-7831; GSK 4182136; GSK-4182136; GSK4182136; VIR 7831; VIR-7831; VIR7831; Monoclonal antibodies against SARS-CoV-2: sotrovimab
Procedure: Biospecimen Collection — Undergo blood and nasal swab sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase I trial studies the process by which sotrovimab is absorbed, distributed, metabolized, and eliminated by the body (pharmacokinetics) in hematopoietic stem cell transplant recipients. Sotrovimab is a monoclonal antibody that may target and bind to a specific protein on SARS-CoV-2 and block its viral attachment and entry into human cells. This may slow the progression of the disease and accelerate recovery, and may potentially provide temporary protection against infection with SARS-CoV-2 in hematopoietic stem cell transplant recipients.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive sotrovimab intravenously (IV) over 30 minutes within 1-7 days prior to the start of pre-transplant conditioning. Patients also undergo blood and nasal swab sample collection throughout the trial.

After completion of study treatment, patients are followed up for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients (or legally authorized representative if applicable) must be capable of understanding and providing a written informed consent
* Patients must be at least 18 years of age, of any gender, race, or ethnicity
* Patients must be undergoing HCT (any donor or stem cell source including autologous or cord blood)
* History of prior transplants are permitted
* History of COVID-19, history of vaccination for SARS-CoV-2, positive polymerase chain reaction (PCR) of a respiratory specimen for SARS-CoV-2 as long as it is not within four weeks from conditioning, or seropositivity for SARS-CoV-2 are permitted
* History of SARS-CoV-2 infection or vaccination of the donor are permitted.
* Post-enrollment vaccination is anticipated and permitted
* Administration of intravenous immunoglobulin therapy (IVIG) before or during the study is permitted

Exclusion Criteria:

* Signs or symptoms of uncontrolled, active infection
* Positive PCR result for SARS-CoV-2 within four weeks of scheduled conditioning
* Pregnant or breastfeeding (this population is generally not cleared for transplant)

  * Pregnancy test is obtained as part of pre-transplant evaluation in women of child-bearing potential at arrival to transplant and again within 7 days of conditioning and will be confirmed as negative by review of the chart
* Previous anaphylaxis or severe hypersensitivity reaction, including angioedema, to a mAb
* Previous reaction to a mAb that required medical attention
* Participants of other clinical studies that preclude the use of other investigational compounds
* Participants who, in the judgment of the investigator, will be unlikely or unable to comply with the requirements of the protocol or unlikely to survive to the end of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alpana Waghmare, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sotrovimab: Patients receive sotrovimab IV over 30 minutes within 1-7 days prior to the start of pre-transplant conditioning. Patients complete questionnaires, blood sample, and nasal swab collections throughout course of trial.
Period: Overall Study
Arm/Group | Sotrovimab
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sotrovimab
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Diagnosis [Count of Participants; unit: Participants]
  Acute leukemia | 5
  T-LGL | 1
  MDS | 5
  MPN (CMML, MF) | 3
  Lymphoma | 3
  Multiple myeloma | 3
Conditioning regimen [Count of Participants; unit: Participants] — Conditioning regimens are determined by clinical teams. Data is collected through chart review. Abbreviations: Bu, busulfan; CLAG-M, cladribine + cytarabine + granulocyte colony-stimulating factor + mitoxantrone; CMML, chronic myelomonocytic leukemia; Cy, cyclophosphamide; Flu, fludarabine; MDS, myelodysplastic syndrome; Mel, melphalan; MF, myelofibrosis; MPN, myeloproliferative neoplasm; TBI, total body irradiation; T-LGL, T-cell large granular lymphocytic leukemia; Treo, treosulfan.
  Participants
    Mel | 3
    Flu/Mel | 2
    Flu/Treo | 1
    Flu/TBI | 3
    Bu/Cy | 1
    Flu/Mel/TBI | 5
    Flu/Cy/TBI | 1
    Bu/Cy/Thiotepa | 1
    Bu/Cy/Thiotepa/Palifermin | 1
    Flu/Cy/Thiotepa/TBI | 1
    CLAG-M/TBI | 1
Type of transplant [Count of Participants; unit: Participants]
  Allogeneic matched unrelated | 8
  Allogeneic matched related | 4
  Allogeneic mismatched unrelated | 1
  Allogeneic cord blood | 2
  Autologous | 5

OUTCOME MEASURES:

1. Primary Outcome: Half-life of Sotrovimab (VIR-7831) Post-transplant
Description: Will use descriptive statistics of model estimation from population pharmacokinetic model. Levels of VIR-7831 can be measured using an idiotypic antibody assay that is not affected by COVID-19 infection or vaccination.
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sotrovimab
Number analyzed (Participants) | 20
Days | 51.14 (18.59)

2. Primary Outcome: Neutralizing Antibody Titers
Description: Will be calculated by a one-phase exponential decay model. Will compare fold-changes in antibody titers by normalizing to pre-transplant levels for each subject. Data analysis was not performed.
Time Frame: Up to 24 weeks
Population: Neutralization assays were not performed, thus no data was collected.
Arm/Group | Sotrovimab
Number analyzed (Participants) | 0

3. Secondary Outcome: Half-life of VIR-7831 in Matched vs Mismatched Donors
Description: Comparisons will be tested using a t-test. Levels of VIR-7831 can be measured using an idiotypic antibody assay that is not affected by COVID-19 infection or vaccination.
Time Frame: Up to 24 weeks
Population: There was only 1 participant in the mismatched group, therefore, sample size was too small to calculate and compare mean or median half-lives between groups. Thus, half-life data was not collected on these groups.
Arm/Group | Sotrovimab
Number analyzed (Participants) | 0

4. Secondary Outcome: Half-life of VIR-7831 in Autologous vs Allogeneic HCT
Description: as for outcome 3
Time Frame: Up to 24 weeks
Population: Two different groups were analyzed based on transplant type. The number of participants in each subgroup will add up to the total number of participants analyzed.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Sotrovimab
Number analyzed (Participants) | 20
Days
  Half-life in autologous participants: number analyzed (Participants) | 5
  Half-life in autologous participants | 63.9 [51.5 to 75.0]
  Half-life in allogeneic participants: number analyzed (Participants) | 15
  Half-life in allogeneic participants | 49.4 [19.5 to 69.7]

5. Secondary Outcome: VIR-7831 Exposure in Patients With Diarrhea vs no Diarrhea
Description: Sotrovimab exposure to be measured as the area under curve (AUC) of sotrovimab concentration over time in model simulation. Comparisons will be tested using a t-test.
Time Frame: Up to 24 weeks
Population: Three different groups were analyzed based on transplant type and presence of diarrhea. The number of patients in each subgroup will add up to the total number of patients analyzed.
Measure: Mean (Standard Deviation); unit: (AUC) micrograms x day/mL
Arm/Group | Sotrovimab
Number analyzed (Participants) | 20
(AUC) micrograms x day/mL
  Allogeneic HCT with diarrhea: number analyzed (Participants) | 11
  Allogeneic HCT with diarrhea | 2027.48 (348.84)
  Allogeneic HCT without diarrhea: number analyzed (Participants) | 4
  Allogeneic HCT without diarrhea | 3613.94 (392.81)
  Autologous HCT without diarrhea: number analyzed (Participants) | 5
  Autologous HCT without diarrhea | 4146.8 (397.57)

6. Secondary Outcome: VIR-7831 Exposure in Patients With and Without Graft Versus Host Disease
Description: Sotrovimab exposure to be measured as the area under curve (AUC) of sotrovimab concentration over time. Comparisons will be tested using a t-test.
Time Frame: Up to 24 weeks
Population: Three different groups were analyzed based on transplant type and presence of lower GI GVHD. The number of patients in each subgroup will add up to the total number of patients analyzed.
Measure: Mean (Standard Deviation); unit: (AUC) micrograms x day/mL
Arm/Group | Sotrovimab
Number analyzed (Participants) | 20
(AUC) micrograms x day/mL
  Allogeneic HCT with lower GI GVHD: number analyzed (Participants) | 10
  Allogeneic HCT with lower GI GVHD | 1846.97 (315.84)
  Allogeneic HCT without lower GI GVHD: number analyzed (Participants) | 5
  Allogeneic HCT without lower GI GVHD | 3613.94 (392.81)
  Autologous HCT without lower GI GVHD: number analyzed (Participants) | 5
  Autologous HCT without lower GI GVHD | 4146.8 (397.57)

7. Secondary Outcome: Number of Participants With Breakthrough SARS-CoV-2 Acquisition
Description: Will monitor for breakthrough SARS-CoV-2 infection by polymerase chain reaction of fluid collected by nasal swabs.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab
Number analyzed (Participants) | 20
Participants | 3

8. Secondary Outcome: Antibody Clearance Rate From Serum/Plasma
Description: Will compare antibody levels from serum/plasma collected by venipuncture versus self-collected using a TASSO device and fluid from nasal swabs. To do this, will compare rate of antibody clearance on average in study population pharmacokinetic model.
Time Frame: Up to 24 weeks
Population: Only those participants with data available at the specified time points were analyzed. Due to early termination, we did not analyze TASSO samples or nasal swabs, hence there is no TASSO or nasal swab data to report.
  Two different groups were analyzed based on transplant type. The number of patients in each subgroup will add up to the total number of patients analyzed.
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | Sotrovimab
Number analyzed (Participants) | 20
L/day
  Elimination clearance in autologous HCT participants: number analyzed (Participants) | 5
  Elimination clearance in autologous HCT participants | 0.1074 (0.0141)
  Elimination clearance in allogeneic HCT participants: number analyzed (Participants) | 15
  Elimination clearance in allogeneic HCT participants | 0.1462 (0.0479)

9. Secondary Outcome: Number of Participants With Presence of Anti-drug Antibodies From Serum/Plasma
Description: Will monitor for presence of anti-drug antibodies from serum/plasma collected by venipuncture versus self-collected using a TASSO device. Samples were considered either positive or negative for presence of anti-drug antibodies.
Time Frame: At 4 and 24 weeks
Population: Only blood collected by venipuncture was assessed. Blood was rarely collected using the TASSO device due to participants declining TASSO use, sotrovimab deauthorization, and early study termination. Limited blood collection with TASSO device, premature study closure, and lack of funds prevented planned laboratory assays on blood collected with the TASSO device. Thus, no laboratory data is available from TASSO-collected blood and no analysis was performed. Further data collection is not planned.
Measure: Count of Participants; unit: Participants
Groups:
- Venipuncture: Patients receive sotrovimab IV over 30 minutes within 1-7 days prior to the start of pre-transplant conditioning. Patients complete questionnaires, blood sample via venipuncture, and nasal swab collections throughout course of trial.
- TASSO Device: Patients receive sotrovimab IV over 30 minutes within 1-7 days prior to the start of pre-transplant conditioning. Patients complete questionnaires, blood sample via self-collected TASSO device, and nasal swab collections throughout course of trial.
Arm/Group | Venipuncture | TASSO Device
Number analyzed (Participants) | 19 | 0
Participants
  Baseline with positive test results | 0 |
  Week 4 with positive test results: number analyzed (Participants) | 18 | 0
  Week 4 with positive test results | 0 |
  Week 24 with positive test results: number analyzed (Participants) | 17 | 0
  Week 24 with positive test results | 0 |

10. Secondary Outcome: Number of Participants With Adverse Events
Description: Will monitor safety with routine labs as part of standard post-transplant care.
Time Frame: Up to 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab
Number analyzed (Participants) | 20
Participants | 4

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Sotrovimab
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotrovimab (N=20)
Death (Gastrointestinal disorders) | 1 (1) — Gastrointestinal hemorrhage is cause of death. Determined to not be related to investigation product.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotrovimab (N=20)
Hypertension stage 2 (Cardiac disorders) | 2 (2) — Occurred following infusion or day after infusion. Unknown if related to investigation product.
Tingling (Injury, poisoning and procedural complications) | 1 (1) — Tingling of arms and chest during product infusion. Paused infusion and improved without additional intervention. Unknown if related to product infusion.

LIMITATIONS AND CAVEATS:
Limitations due to small sample size: Relatively low precision in estimating covariate effects. Models/data presented focus on GI GVHD as cause of diarrhea; subgroup analysis couldn't be performed to examine whether different pretransplant preparative regimens were associated with increased mAb elimination. Did not perform covariate analysis on varying types of allogeneic HCT.

Study halted prematurely due to emergence of variants with reduced in vitro neutralization to sotrovimab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT05135650/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT05135650/ICF_000.pdf